CLINICAL TRIAL: NCT01979094
Title: General Spinal Arthrodesis and Spinal Arthroplasty Database
Brief Title: Spinal Arthrodesis and Spinal Arthroplasty Database Study
Status: Terminated | Type: Observational
Why Stopped: Process changes. New data base will be activated
Sponsor: Stephanus Viljoen (Other)
Responsible Party: Sponsor-Investigator, Stephanus Viljoen, Assistant Professor, Ohio State University
Organization: Ohio State University (Other)
Other Study IDs: 2013H0104
Record Dates: First submitted 2013-10-24; First posted 2013-11-08 (Estimated); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Spine Condition

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- spinal arthrodesis and/or arthroplasty procedures

SUMMARY:
To collect and organize data into a repository for future research.

DETAILED DESCRIPTION:
To collect and organize data into a repository from the Principal Investigator's (H. Francis Farhadi, MD, PhD) patients who are undergoing spinal arthrodesis and/or spinal arthroplasty procedures at Ohio State University for future research, as yet to be identified. This comprehensive database of patients will allow for gathering of relevant information for potential future research use.

ELIGIBILITY:
Inclusion Criteria:

* Must have had or will undergo a spinal arthrodesis and/or spinal arthroplasty procedure at Ohio State University

Exclusion Criteria:

* N/A

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Spinal arthrodesis and/or spinal arthroplasty can be performed through either anterior, posterior, or lateral approaches for a variety of traumatic, degenerative, or deformity conditions.
Sampling Method: Probability Sample
Enrollment: 1296 (Actual)
Dates: Start 2013-05; Primary Completion 2024-01-04 (Actual); Study Completion 2024-01-04 (Actual)

PRIMARY OUTCOMES:
clinical prospective review- Prospective Database study for future studies | 5 years
  Collecting clinical measurements. Examples of these clinical measurements are the VAS Pain Scale, SF-36, NDI, and ODI.

CONTACTS AND LOCATIONS:
Overall Officials: H. Francis Farhadi, MD, PhD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State Unviersity, Columbus, Ohio, United States